CLINICAL TRIAL: NCT02774538
Title: Agreement Between Oral and Cervical Human Papillomavirus Infection in a French Cohort of Women Infected With Cervical HPV
Brief Title: Agreement Between Oral and Cervical Human Papillomavirus Infection in a French Cohort
Acronym: PAPILLOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-A00594-45
Record Dates: First submitted 2016-05-03; First posted 2016-05-17 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Human Papillomavirus-Related Cervical Carcinoma
Keywords: Cervical HPV infection; Oral HPV infection; Sexually transmitted infection
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Other)
  Interventions: Other: Agreement between oral and cervical HPV infection

INTERVENTIONS:
Other: Agreement between oral and cervical HPV infection — A total of 165 women will have a Pap test and an oral brushing performed on the day of inclusion. Risk factors for oral HPV infection will be defined using a self-administered survey summarizing the demographics and sexual behaviors.
  A second oral brushing up to 18 months will be performed during a standard follow-up visit.

SUMMARY:
Human papillomaviruses (HPVs) are the most common of sexually transmitted viral agents and they are associated with genital and oral diseases.

Agreement between cervical and oral HPV infection has been described from a small group of patient. Our study, performed on a greater number of patients, will provide a good estimation of this link, between cervical and oral infection, in a French population of women with a primary cervical HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proven of cervical intraepithelial neoplasia or carcinoma in situ (CIS) or invasive cervical cancer or a Pap smear on which at least one HPV has been detected
* Patients not vaccinated against HPV
* Age >18 years
* EOCG performance status ≤ 3
* Patient must be affiliated to a social security system
* Ability to provide written informed consent patient's legal capacity to consent to study participation and to understand and comply with the requirements of the study

Exclusion Criteria:

* Patients vaccinated against HPV
* Pregnant woman over 10 weeks
* Patient who underwent head and neck radiotherapy dating less than one year
* Patients deprived of liberty or under supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Agreement between oral and cervical HPV infection | up to 6 months
  Agreement between oral and cervical HPV infection is defined by the presence of at least one identical genotype HPV in both sites in the same wife. All genotypes found in the oral and cervical area will be considered.

SECONDARY OUTCOMES:
Agreement between full and partial oral and cervical HPV genotypes | up to 6 months
  Agreement between oral and cervical HPV genotypes is considered as complete if the same HPV genotypes were detected on both sites. Agreement between oral and cervical HPV genotypes is considered as partial when at least one but not all HPV genotypes were detected at both sites.
Proportion of women with oral HPV infection in women with primary cervical HPV infection | up to 6 months
Proportion of women with oral high risk HPV infection | up to 6 months
Description of all HPV genotypes found in women with HPV infection at both sites | up to 6 months
  All genotypes found in the oral and cervical area will be described.
Oral HPV risk factors | up to 6 months
  The following oral HPV risk factors will be analyzed: smoking, regular alcohol consumption, number of sexual partners, sexual risk behaviors.
Persistence and clearance of oral HPV infection | up to 18 months
  The persistence of HPV infection will be defined by the detection of the same genotype of oral HPV between the two tests.
  The clearance of HPV infection will be defined by a positive oral HPV infection at baseline and a negative oral HPV infection up to 18 months.
Frequency of newly positive women with oral HPV infection | up to 18 months
  Women with no HPV infection at baseline and positive HPV infection at 18 months will be considered as newly positive women.

CONTACTS AND LOCATIONS:
Overall Officials: GUILLET Julie, Dr, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (4):
- France (4):
  - Hôpital Nord Franche-Comté, Belfort
  - CHRU Besançon, Besançon
  - Maternité Régionale Universitaire de Nancy, Nancy
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No